CLINICAL TRIAL: NCT00673387
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Examine the Safety, Tolerability, and Effect on Body Weight of Metreleptin Administered in Conjunction With Pramlintide in Obese and Overweight Subjects.
Brief Title: Study to Examine Safety, Tolerability, and Effect on Body Weight of Metreleptin Administered in Conjunction With Pramlintide in Obese and Overweight Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: DFA102
Record Dates: First submitted 2008-05-06; First posted 2008-05-07 (Estimated); Results first posted 2013-11-14 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-03

CONDITIONS: Overweight; Obesity
Keywords: overweight; obesity; pramlintide; metreleptin; Amylin
MeSH Terms: conditions — Overweight; Obesity | interventions — pramlintide; metreleptin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Placebo-P + Placebo-M (Placebo Comparator): Placebo matched to pramlintide BID plus placebo matched to metreleptin BID
  Interventions: Drug: placebo-P; Drug: placebo-M
- Pramlintide 360 mcg + Placebo-M (Experimental): 360 mcg pramlintide given twice per day (BID) plus Placebo matched to Metreleptin given BID
  Interventions: Drug: pramlintide acetate; Drug: placebo-M
- Placebo-P + Metreleptin 5.0 mg (Experimental): Placebo matched to pramlintide BID plus metreleptin 5.0 mg BID
  Interventions: Drug: metreleptin; Drug: placebo-P
- Pramlintide 180 mcg + Metreleptin 2.5 mg (Experimental): Pramlintide 180 mcg BID plus Metreleptin 2.5 mg BID
  Interventions: Drug: pramlintide acetate; Drug: metreleptin
- Pramlintide 180 mcg + Metreleptin 5.0 mg (Experimental): Pramlintide 180 mcg BID plus Metreleptin 5.0 mg BID
  Interventions: Drug: pramlintide acetate; Drug: metreleptin
- Pramlintide 360 mcg + Metreleptin 1.25 mg (Experimental): Pramlintide 360 mcg BID plus Metreleptin 1.25 mg BID
  Interventions: Drug: pramlintide acetate; Drug: metreleptin
- Pramlintide 360 mcg + Metreleptin 2.5 mg (Experimental): Pramlintide 360 mcg BID plus Metreleptin 2.5 mg BID
  Interventions: Drug: pramlintide acetate; Drug: metreleptin
- Pramlintide 360 mcg + Metreleptin 5.0 mg (Experimental): Pramlintide 360 mcg BID plus Metreleptin 5.0 mg BID
  Interventions: Drug: pramlintide acetate; Drug: metreleptin

INTERVENTIONS:
Drug: pramlintide acetate — subcutaneous injection, twice a day
  Other Names: Smylin
  Arms: Pramlintide 180 mcg + Metreleptin 2.5 mg; Pramlintide 180 mcg + Metreleptin 5.0 mg; Pramlintide 360 mcg + Metreleptin 1.25 mg; Pramlintide 360 mcg + Metreleptin 2.5 mg; Pramlintide 360 mcg + Metreleptin 5.0 mg; Pramlintide 360 mcg + Placebo-M
Drug: metreleptin — subcutaneous injection, twice a day
  Arms: Placebo-P + Metreleptin 5.0 mg; Pramlintide 180 mcg + Metreleptin 2.5 mg; Pramlintide 180 mcg + Metreleptin 5.0 mg; Pramlintide 360 mcg + Metreleptin 1.25 mg; Pramlintide 360 mcg + Metreleptin 2.5 mg; Pramlintide 360 mcg + Metreleptin 5.0 mg
Drug: placebo-P — subcutaneous injection, twice a day
  Other Names: Placebo matched to pramlintide
  Arms: Placebo-P + Metreleptin 5.0 mg; Placebo-P + Placebo-M
Drug: placebo-M — subcutaneous injection, twice a day
  Other Names: Placebo matched to Metreleptin
  Arms: Placebo-P + Placebo-M; Pramlintide 360 mcg + Placebo-M

SUMMARY:
A randomized, double-blind, placebo-controlled, dose-ranging study to examine the safety, tolerability and effect on body weight of a range of doses of metreleptin and pramlintide, each administered by a separate subcutaneous (SC) injection in obese and overweight subjects.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years old.
* Is obese (Body Mass Index [BMI]>=30kg/m^2 and <=35kg/m^2); or overweight (BMI>=27kg/m^2 and <30kg/m^2.
* Has stable body weight, i.e., not varying by >3% within 3 months prior to study.
* Has not been treated over the past 3 months or is currently treated with any of the following medications: Oral contraceptives (female subjects); Hormone replacement therapy (female subjects); Metformin for the treatment of polycystic ovary syndrome (female subjects); Antihypertensive agents; Lipid-lowering agents; Thyroid replacement therapy; selective serotonin reuptake inhibitors (SSRIs).
* Is comfortable with having repeated telephone contacts with a lifestyle counselor during the study.
* Is a nonsmoker (has not smoked for at least 6 months prior to the study).

Exclusion Criteria:

* Has a medical history (e.g., morbid childhood obesity) and/or physical characteristics suggestive of genetic obesity or syndromatic obesity (e.g., Prader-Willi syndrome, Bardet-Biedl syndrome).
* Is currently enrolled or plans to enroll in a diet, weight loss, or exercise program with the specific intent of losing weight (subjects who have been following an exercise regimen resulting in stable weight maintenance for at least 2 months prior to enrollment are eligible for study inclusion)
* Has been treated over the past 2 months, is currently treated, or is expected to require or undergo treatment with *antiobesity agents (prescription or over-the-counter), *antipsychotic agents, *antiepileptic agents, *antidepressant agents, *drugs that directly affect gastrointestinal motility, *antidiabetic medications.
* Has previously received treatment with metreleptin or pramlintide in a clinical study or has received prior treatment with pramlintide (SYMLIN®).
* Has received any investigational drug within 30 days or within a period corresponding to 5 half-lives of that drug, whichever is greater, prior to this study starting.
* Has had a major surgery or a blood transfusion, or has donated blood over the past 2 months or is planning to donate blood during the study.
* Has had liposuction, abdominoplasty, or similar procedure over the past year or is planning to have such a procedure during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 636 (Actual)
Dates: Start 2008-04; Primary Completion 2009-04 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vice President Research and Development, MD, Study Director — Amylin Pharmaceuticals, LLC.
Locations (36):
- United States (36):
  - Research Site, Birmingham, Alabama
  - Research Site, Chandler, Arizona
  - Research Site, Santa Rosa, California
  - Research Site, Walnut Creek, California
  - Research Site, Denver, Colorado
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Pembrook Pines, Florida
  - Research Site, Plantation, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Springfield, Illinois
  - Research Site, Overland Park, Kansas
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Auburn, Maine
  - Research Site, Boston, Massachusetts
  - Research Site, Edina, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Butte, Montana
  - Research Site, New York, New York
  - Research Site, Statesville, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Eugene, Oregon
  - Research Site, Medford, Oregon
  - Research Site, Anderson, South Carolina
  - Research Site, Greer, South Carolina
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Norfolk, Virginia
  - Research Site, Belingham, Washington
  - Research Site, Olympia, Washington

REFERENCES:
- [Derived] Chan JL, Koda J, Heilig JS, Cochran EK, Gorden P, Oral EA, Brown RJ. Immunogenicity associated with metreleptin treatment in patients with obesity or lipodystrophy. Clin Endocrinol (Oxf). 2016 Jul;85(1):137-49. doi: 10.1111/cen.12980. Epub 2016 Feb 2. PMID 26589105

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant dosed/lead in: 06 May 2008; last participant's final visit: 07 April 2009. Study conducted in 42 clinics in participants who were either obese (body mass index (BMI) greater than, equal to (>=) 30 kg/m^2 and less than equal to (<=) 45 kg/m^2) or overweight (>= 27 kg/m^2 and < 30 kg/m^2).
Pre-assignment Details: Participants enrolled, not randomized /treated (28): withdrew consent (10), adverse event (1), investigator decision (7), protocol violation (4), lost to follow up (5), administrative (1). 1 Week Lead-in Period: all arms received placebo matched to metreleptin and matched to pramlintide, BID (single blind); 28 week double blind Treatment Period.
Groups:
- Placebo: Self administered twice a day (BID) for 28 weeks, subcutaneous (SC) placebo matched to pramlintide (Placebo-P) plus SC placebo matched to metreleptin (Placebo-M).
- Pramlintide 360 mcg: Self administered BID for 28 weeks, SC 360 mcg pramlintide acetate plus SC Placebo matched to Metreleptin (Placebo-M). The first week of the 28 weeks started with a lower pramlintide dose (180 mcg) in a blinded fashion (using 2 different concentrations of pramlintide so the dose change was not apparent to the participant).
- Metreleptin 5.0 mg: Self administered BID for 28 weeks, SC metreleptin 5.0 mg plus SC Placebo matched to pramlintide (Placebo-P).
- Pramlintide 180 mcg + Metreleptin 2.5 mg: Self administered BID for 28 weeks, SC Pramlintide 180 mcg plus SC Metreleptin 2.5 mg.
- Pramlintide 180 mcg + Metreleptin 5.0 mg: Self administered BID for 28 weeks, SC Pramlintide 180 mcg plus SC Metreleptin 5.0 mg
- Pramlintide 360 mcg + Metreleptin 1.25 mg: Self administered BID for 28 weeks, SC Pramlintide 360 mcg plus SC Metreleptin 1.25 mg. The first week of the 28 weeks started with a lower pramlintide dose (180 mcg) in a blinded fashion (using 2 different concentrations of pramlintide so the dose change was not apparent to the participant).
- Pramlintide 360 mcg + Metreleptin 2.5 mg: Self administered BID for 28 weeks, SC Pramlintide 360 mcg plus SC Metreleptin 2.5 mg. The first week of the 28 weeks started with a lower pramlintide dose (180 mcg) in a blinded fashion (using 2 different concentrations of pramlintide so the dose change was not apparent to the participant).
- Pramlintide 360 mcg + Metreleptin 5.0 mg: Self administered BID for 28 weeks, SC Pramlintide 360 mcg plus SC Metreleptin 5.0 mg. The first week of the 28 weeks started with a lower pramlintide dose (180 mcg) in a blinded fashion (using 2 different concentrations of pramlintide so the dose change was not apparent to the participant).
Period: Overall Study
Arm/Group | Placebo | Pramlintide 360 mcg | Metreleptin 5.0 mg | Pramlintide 180 mcg + Metreleptin 2.5 mg | Pramlintide 180 mcg + Metreleptin 5.0 mg | Pramlintide 360 mcg + Metreleptin 1.25 mg | Pramlintide 360 mcg + Metreleptin 2.5 mg | Pramlintide 360 mcg + Metreleptin 5.0 mg
Started | 75 | 77 | 72 | 75 | 78 | 78 | 78 | 75
Completed | 46 | 54 | 41 | 49 | 48 | 44 | 48 | 40
Not Completed | 29 | 23 | 31 | 26 | 30 | 34 | 30 | 35
Not completed — Withdrawal by Subject | 15 | 16 | 20 | 16 | 18 | 21 | 15 | 21
Not completed — Adverse Event | 3 | 1 | 5 | 2 | 6 | 2 | 5 | 5
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 1
Not completed — Protocol Violation | 3 | 0 | 1 | 2 | 0 | 1 | 1 | 3
Not completed — Lost to Follow-up | 8 | 6 | 5 | 6 | 6 | 5 | 8 | 5

BASELINE CHARACTERISTICS:
Population: Intent to treat population. All participants randomized to a treatment and received at least 1 dose. Drug Randomization stratified:sex,3 categories baseline BMI (12 arms); 3 treatment arms combined for summaries as single placebo treatment group; 3 combined for summaries as single pramlintide monotherapy treatment group (total:8 treatment groups).
Groups:
- Placebo: Self administered BID for 28 weeks, SC placebo matched to pramlintide (Placebo-P) plus SC placebo matched to metreleptin (Placebo-M).
- Total: Total of all reporting groups
Arm/Group | Placebo | Pramlintide 360 mcg | Metreleptin 5.0 mg | Pramlintide 180 mcg + Metreleptin 2.5 mg | Pramlintide 180 mcg + Metreleptin 5.0 mg | Pramlintide 360 mcg + Metreleptin 1.25 mg | Pramlintide 360 mcg + Metreleptin 2.5 mg | Pramlintide 360 mcg + Metreleptin 5.0 mg | Total
Number analyzed (Participants) | 75 | 77 | 72 | 75 | 78 | 78 | 78 | 75 | 608
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.9 (11.35) | 42.0 (11.42) | 45.9 (10.92) | 45.8 (10.80) | 46.8 (10.54) | 44.4 (10.87) | 45.2 (10.07) | 44.7 (11.32) | 44.6 (10.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 54 | 53 | 53 | 54 | 54 | 55 | 52 | 428
  Male | 22 | 23 | 19 | 22 | 24 | 24 | 23 | 23 | 180
Region of Enrollment [Number; unit: participants]
  United States | 75 | 77 | 72 | 75 | 78 | 78 | 78 | 75 | 608
Body Mass Index [Mean (Standard Deviation); unit: (kg/m^2)] — Body Mass Index (BMI)calculated using baseline weight and height; BMI = kg body weight/meters of height^2. Weight, height measured on Day 1. If Day 1 value missing or value obtained after the first dose, the last available value prior to Day 1 was used.
  (kg/m^2) | 36.88 (4.473) | 36.93 (4.389) | 36.62 (4.478) | 36.88 (4.336) | 36.65 (4.379) | 36.80 (4.260) | 36.96 (4.406) | 36.68 (4.504) | 36.80 (4.379)

OUTCOME MEASURES:

1. Primary Outcome: Least Squares (LS) Mean Percent Change in Body Weight From Baseline to Week 28 - Evaluable Population
Description: Body weight was measured in kilogram (kg). Baseline is defined as Day 1. If Day 1 was missing or after the first dose date of randomized treatment, the last available value prior to Day 1 was used. Drug Randomization stratified by sex and 3 categories baseline BMI (12 arms); 3 treatment arms combined for summaries as single placebo treatment group; 3 combined for summaries as single pramlintide monotherapy treatment group (total: 8 treatment groups).
Time Frame: Baseline to Week 28
Population: Evaluable population includes all intent to treat participants (received at least one dose of randomized treatment) who had adequate exposure to treatment and complied with the protocol as assessed prior to database lock and unblinding.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change in kg
Arm/Group | Placebo | Pramlintide 360 mcg | Metreleptin 5.0 mg | Pramlintide 180 mcg + Metreleptin 2.5 mg | Pramlintide 180 mcg + Metreleptin 5.0 mg | Pramlintide 360 mcg + Metreleptin 1.25 mg | Pramlintide 360 mcg + Metreleptin 2.5 mg | Pramlintide 360 mcg + Metreleptin 5.0 mg
Number analyzed (Participants) | 47 | 51 | 41 | 47 | 46 | 45 | 45 | 38
Percentage change in kg | -2.01 [-3.76 to -0.26] | -5.47 [-7.19 to -3.76] | -5.83 [-7.72 to -3.95] | -6.85 [-8.61 to -5.08] | -6.61 [-8.41 to -4.82] | -6.39 [-8.18 to -4.59] | -6.98 [-8.79 to -5.17] | -7.02 [-8.94 to -5.10]
Statistical Analysis 1: Comparison: Placebo vs Pramlintide 180 mcg + Metreleptin 2.5 mg; When multiplicity not considered, sample size of 50 participants per arm (after dropouts) was considered adequate to detect a difference of 4.5% in mean body weight change from baseline to Week 28 between one effective pramlintide + metreleptin combination treatment group versus the placebo, Pramlintide 360 mcg BID + Placebo-M, or Metreleptin 5.0 mg BID + Placebo-P treatment arms with approximately 90% power, assuming a common within-treatment standard deviation of 6.858%; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — unadjusted for multiple comparisons; significance level of 0.0492 based on the Haybittle-Peto Criterion
Statistical Analysis 2: Comparison: Placebo vs Pramlintide 180 mcg + Metreleptin 5.0 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0002, t-test, 2 sided — unadjusted for multiple comparisons; significance level of 0.0492 based on the Haybittle-Peto Criterion
Statistical Analysis 3: Comparison: Placebo vs Pramlintide 360 mcg + Metreleptin 1.25 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0004, t-test, 2 sided — unadjusted for multiple comparisons; significance level of 0.0492 based on the Haybittle-Peto Criterion
Statistical Analysis 4: Comparison: Placebo vs Pramlintide 360 mcg + Metreleptin 2.5 mg; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — unadjusted for multiple comparisons; significance level of 0.0492 based on the Haybittle-Peto Criterion
Statistical Analysis 5: Comparison: Placebo vs Pramlintide 360 mcg + Metreleptin 5.0 mg; Test type: Superiority or Other; p = 0.0001, t-test, 2 sided — unadjusted for multiple comparisons; significance level of 0.0492 based on the Haybittle-Peto Criterion
Statistical Analysis 6: Comparison: Pramlintide 360 mcg vs Pramlintide 180 mcg + Metreleptin 2.5 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2510, t-test, 2 sided — unadjusted for multiple comparisons; significance level of 0.0492 based on the Haybittle-Peto Criterion
Statistical Analysis 7: Comparison: Pramlintide 360 mcg vs Pramlintide 180 mcg + Metreleptin 5.0 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3433, t-test, 2 sided — unadjusted for multiple comparisons; significance level of 0.0492 based on the Haybittle-Peto Criterion
Statistical Analysis 8: Comparison: Pramlintide 360 mcg vs Pramlintide 360 mcg + Metreleptin 1.25 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4503, t-test, 2 sided — unadjusted for multiple comparisons; significance level of 0.0492 based on the Haybittle-Peto Criterion
Statistical Analysis 9: Comparison: Pramlintide 360 mcg vs Pramlintide 360 mcg + Metreleptin 2.5 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2122, t-test, 2 sided — unadjusted for multiple comparisons; significance level of 0.0492 based on the Haybittle-Peto Criterion
Statistical Analysis 10: Comparison: Pramlintide 360 mcg vs Pramlintide 360 mcg + Metreleptin 5.0 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2232, t-test, 2 sided — unadjusted for multiple comparisons; significance level of 0.0492 based on the Haybittle-Peto Criterion
Statistical Analysis 11: Comparison: Metreleptin 5.0 mg vs Pramlintide 180 mcg + Metreleptin 2.5 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4207, t-test, 2 sided — unadjusted for multiple comparisons; significance level of 0.0492 based on the Haybittle-Peto Criterion
Statistical Analysis 12: Comparison: Metreleptin 5.0 mg vs Pramlintide 180 mcg + Metreleptin 5.0 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5375, t-test, 2 sided — unadjusted for multiple comparisons; significance level of 0.0492 based on the Haybittle-Peto Criterion
Statistical Analysis 13: Comparison: Metreleptin 5.0 mg vs Pramlintide 360 mcg + Metreleptin 1.25 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6633, t-test, 2 sided — unadjusted for multiple comparisons; significance level of 0.0492 based on the Haybittle-Peto Criterion
Statistical Analysis 14: Comparison: Metreleptin 5.0 mg vs Pramlintide 360 mcg + Metreleptin 2.5 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3667, t-test, 2 sided — unadjusted for multiple comparisons; significance level of 0.0492 based on the Haybittle-Peto Criterion
Statistical Analysis 15: Comparison: Metreleptin 5.0 mg vs Pramlintide 360 mcg + Metreleptin 5.0 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3720, t-test, 2 sided — unadjusted for multiple comparisons; significance level of 0.0492 based on the Haybittle-Peto Criterion

2. Secondary Outcome: Number of Participants Achieving at Least 5% and at Least 10% Body Weight Loss From Baseline to Week 28 - Evaluable Population
Description: Baseline refers to Day 1. If Day 1 value is missing or after the first dose date of randomized study medication, the last available value on or prior to Day 1 is used.
Time Frame: Baseline to Week 28
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | Pramlintide 360 mcg | Metreleptin 5.0 mg | Pramlintide 180 mcg + Metreleptin 2.5 mg | Pramlintide 180 mcg + Metreleptin 5.0 mg | Pramlintide 360 mcg + Metreleptin 1.25 mg | Pramlintide 360 mcg + Metreleptin 2.5 mg | Pramlintide 360 mcg + Metreleptin 5.0 mg
Number analyzed (Participants) | 47 | 51 | 41 | 47 | 46 | 45 | 45 | 38
participants
  Weight Loss >=5% | 10 | 27 | 18 | 27 | 27 | 23 | 29 | 25
  Weight Loss >=5% and <10% | 7 | 14 | 6 | 14 | 15 | 15 | 15 | 12
  Weight Loss >=10% | 3 | 13 | 12 | 13 | 12 | 8 | 14 | 13
  Weight Gain | 17 | 7 | 7 | 4 | 8 | 5 | 4 | 3
  No Weight Change or Weight Loss <5% | 20 | 17 | 16 | 16 | 11 | 17 | 12 | 10

3. Secondary Outcome: Mean Absolute Change From Baseline to Weeks 4, 12, 28 in Mean Trough Concentration of Total Leptin - Evaluable Population
Description: Mean fasting plasma total leptin concentration (nanograms per milliliter; ng/mL) change from baseline over time by pooled metreleptin dose (sex, baseline BMI category, and baseline value). Baseline defined as Day 1. If Day 1 value is missing or after the first dose date of randomized study medication, the last available value on or prior to Day 1 is used. Evaluable population: all participants who received at least one dose of randomized treatment, had adequate exposure to treatment and complied with the protocol as assessed prior to database lock and unblinding. Leptin concentrations measured using a validated immunoenzymetric assay utilizing polyclonal capture antibody, monoclonal detection antibody, and colorimetric readout by Amylin Pharmaceuticals, Inc.
Time Frame: Baseline to Week 28
Population: Number analyzed (n) at baseline above. Week 4: n=41 45,46, 45, 45, 38; Week 8: n=41,45,46,44,45,37; Week 12: n=41, 46, 46, 45,45,38; Week 16: n=41,47,46,45,45,38; Week 20: n=41, 45,45,45,45,38; Week 24: n=40, 43, 46, 42, 44,38; Week 28: n=41, 45, 45, 44, 43, 36. Leptin concentration for placebo and pramlintide plus placebo groups not presented.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Metreleptin 5.0 mg | Pramlintide 180 mcg + Metreleptin 2.5 mg | Pramlintide 180 mcg + Metreleptin 5.0 mg | Pramlintide 360 mcg + Metreleptin 1.25 mg | Pramlintide 360 mcg + Metreleptin 2.5 mg | Pramlintide 360 mcg + Metreleptin 5.0 mg
Number analyzed (Participants) | 41 | 47 | 46 | 45 | 45 | 38
ng/mL
  Change from baseline at Week 4 | 53.26 (64.542) | 31.00 (73.953) | 47.82 (76.469) | -2.36 (16.918) | 14.66 (48.212) | 49.16 (70.881)
  Change from baseline at Week 12 | 386.48 (408.472) | 167.62 (147.512) | 353.61 (265.727) | 53.76 (68.627) | 165.65 (173.851) | 399.74 (378.120)
  Change from baseline at Week 28 | 557.22 (604.617) | 373.64 (465.511) | 487.17 (625.071) | 105.96 (143.680) | 266.02 (210.412) | 393.06 (381.428)

4. Secondary Outcome: LS Mean Absolute Change in Body Weight From Baseline to Weeks 4, 12, and 28 - Evaluable Population
Description: Least Squares (LS) mean absolute change in Body weight was measured in kilograms (kg). Baseline is defined as Day 1. If Day 1 was missing or after the first dose date of randomized treatment, the last available value prior to Day 1 was used.
Time Frame: Baseline to Week 28
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Placebo | Pramlintide 360 mcg | Metreleptin 5.0 mg | Pramlintide 180 mcg + Metreleptin 2.5 mg | Pramlintide 180 mcg + Metreleptin 5.0 mg | Pramlintide 360 mcg + Metreleptin 1.25 mg | Pramlintide 360 mcg + Metreleptin 2.5 mg | Pramlintide 360 mcg + Metreleptin 5.0 mg
Number analyzed (Participants) | 47 | 51 | 41 | 47 | 46 | 45 | 45 | 38
kg
  Change at Week 4 | -1.81 [-2.38 to -1.24] | -2.85 [-3.41 to -2.29] | -2.54 [-3.15 to -1.92] | -2.94 [-3.51 to -2.36] | -2.40 [-2.99 to -1.82] | -2.62 [-3.21 to -2.04] | -3.21 [-3.80 to -2.62] | -3.32 [-3.95 to -2.69]
  Change at Week 12 | -3.39 [-4.50 to -2.28] | -4.90 [-5.97 to -3.83] | -5.13 [-6.31 to -3.95] | -5.52 [-6.63 to -4.42] | -4.53 [-5.65 to -4.41] | -5.52 [-6.64 to -4.40] | -5.88 [-7.02 to -4.75] | -6.12 [-7.32 to -4.92]
  Change at Week 28 | -2.04 [-3.82 to -0.26] | -5.66 [-7.40 to -3.92] | -6.18 [-8.10 to -4.27] | -6.96 [-8.75 to -5.17] | -6.55 [-8.38 to -4.72] | -6.38 [-8.20 to -4.56] | -7.18 [-9.03 to -5.34] | -6.97 [-8.92 to -5.02]

5. Secondary Outcome: LS Mean Change in Waist Circumference From Baseline to Week 12 and Week 28 - Evaluable Population
Description: Waist circumference was measured at baseline (Day 1), Weeks 12, 28 (or at early termination) in centimeters (cm).
Time Frame: Baseline to Weeks 12 and Week 28
Population: Participants who received at least 1 dose of randomized treatment and who had adequate exposure to treatment and complied with the protocol as assessed prior to database lock/unblinding. Numbers (n) analyzed Week 12 n=45,51,41,47,45,45,45,38 in each treatment group respectively; Week 28 n= 44, 51, 41, 46, 45, 44, 43, 38 in each group, respectively.
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Placebo | Pramlintide 360 mcg | Metreleptin 5.0 mg | Pramlintide 180 mcg + Metreleptin 2.5 mg | Pramlintide 180 mcg + Metreleptin 5.0 mg | Pramlintide 360 mcg + Metreleptin 1.25 mg | Pramlintide 360 mcg + Metreleptin 2.5 mg | Pramlintide 360 mcg + Metreleptin 5.0 mg
Number analyzed (Participants) | 45 | 51 | 41 | 47 | 45 | 45 | 45 | 38
cm
  Change at Week 12 | -3.03 (0.851) | -3.40 (0.799) | -3.41 (0.895) | -4.91 (0.846) | -4.29 (0.876) | -3.32 (0.853) | -4.63 (0.855) | -5.23 (0.916)
  Change at Week 28 | -2.54 (1.038) | -3.95 (0.965) | -3.86 (1.081) | -5.48 (1.032) | -5.75 (1.058) | -4.70 (1.043) | -5.52 (1.057) | -6.53 (1.107)
Statistical Analysis 1: Comparison: Placebo vs Pramlintide 180 mcg + Metreleptin 2.5 mg; Change at Week 28 based on a general linear model with factors for treatment group, sex, baseline BMI category, and baseline value as a covariate; Test type: Superiority or Other; p = 0.0404, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo vs Pramlintide 180 mcg + Metreleptin 5.0 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0265, t-test, 2 sided
Statistical Analysis 3: Comparison: Placebo vs Pramlintide 360 mcg + Metreleptin 1.25 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.1357, t-test, 2 sided
Statistical Analysis 4: Comparison: Placebo vs Pramlintide 360 mcg + Metreleptin 2.5 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0409, t-test, 2 sided
Statistical Analysis 5: Comparison: Placebo vs Pramlintide 360 mcg + Metreleptin 5.0 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0082, t-test, 2 sided

6. Secondary Outcome: Geometric Mean of the Total Area Under the Concentration Time Curve (AUC) From Time 0 to Last Quantifiable Concentration (Tlast) for Pramlintide at Weeks 4 and 24 - Evaluable Population Receiving Pramlintide
Description: Assessment of AUC was over a period of 2 hours following pramlintide administration. AUC (0 to time of last quantifiable concentration (-tlast). For AUC calculation, concentration at -5 min will be considered as 0 h concentration if quantifiable, otherwise, t=0 h. AUC measured as picograms*hour/milliliter (pg*h/mL). Pramlintide concentrations measured using a colorimetric immunoenzymetric assay employing monoclonal antibodies against pramlintide for both capture and detection.
Time Frame: Week 4 and Week 24
Population: Evaluable population: participants received at least one dose of randomized treatment, had adequate exposure to treatment and complied with the protocol as assessed prior to database lock and unblinding. Number (n) analyzed at Week 4:n=46, 40,41, 40,40,33 in each arm respectively;Week 24:n=48, 38, 44, 40, 35, 36.
Measure: Geometric Mean (Standard Error); unit: pg*h/mL
Groups:
- Pramlintide 360 mcg + Placebo-M: Self administered BID for 28 weeks, SC 360 mcg pramlintide acetate plus SC Placebo matched to Metreleptin (Placebo-M). The first week of the 28 weeks started with a lower pramlintide dose (180 mcg) in a blinded fashion (using 2 different concentrations of pramlintide so the dose change was not apparent to the participant).
Arm/Group | Pramlintide 360 mcg + Placebo-M | Pramlintide 180 mcg + Metreleptin 2.5 mg | Pramlintide 180 mcg + Metreleptin 5.0 mg | Pramlintide 360 mcg + Metreleptin 1.25 mg | Pramlintide 360 mcg + Metreleptin 2.5 mg | Pramlintide 360 mcg + Metreleptin 5.0 mg
Number analyzed (Participants) | 48 | 40 | 44 | 40 | 40 | 36
pg*h/mL
  Week 4 AUC (0-tlast) | 1862.5 (176.83) | 878.8 (87.34) | 967.5 (68.59) | 1788.2 (165.32) | 1920.1 (143.54) | 2060.4 (168.92)
  Week 24 AUC (0-tlast) | 1968.4 (135.60) | 1033.8 (102.19) | 953.7 (76.19) | 1536.3 (103.90) | 1990.2 (160.49) | 1915.3 (158.77)

7. Secondary Outcome: Geometric Mean of AUC From Time 0 to Infinity for Pramlintide at Weeks 4 and 24 - Evaluable Population Treated With Pramlintide
Description: Assessment of AUC was over a period of 2 hours following pramlintide administration. Area under the concentration curve (AUC) time 0 to infinity (-inf). For AUC calculations, concentration at -5 min will be considered as 0 h concentration if quantifiable. AUC measured in picograms*hour/milliliter (pg*h/mL).
Time Frame: Weeks 4 and 24
Population: Evaluable population: participants received at least one dose of randomized treatment, had adequate exposure to treatment and complied with the protocol as assessed prior to database lock and unblinding. Number (n) analyzed at Week 4: n=39,36,37,36,35,31 in each arm, respectively; Week 24 n=46, 35, 42, 39, 33, 35 in each arm, respectively.
Measure: Geometric Mean (Standard Error); unit: pg*h/mL
Arm/Group | Pramlintide 360 mcg + Placebo-M | Pramlintide 180 mcg + Metreleptin 2.5 mg | Pramlintide 180 mcg + Metreleptin 5.0 mg | Pramlintide 360 mcg + Metreleptin 1.25 mg | Pramlintide 360 mcg + Metreleptin 2.5 mg | Pramlintide 360 mcg + Metreleptin 5.0 mg
Number analyzed (Participants) | 46 | 36 | 42 | 39 | 35 | 35
pg*h/mL
  Week 4 AUC (0-inf) | 2662.7 (230.34) | 989.3 (96.05) | 1240.7 (106.08) | 2159.0 (238.45) | 2311.3 (211.63) | 2511.4 (241.16)
  Week 24 AUC (0-inf) | 2499.5 (215.51) | 1175.1 (116.89) | 1216.7 (102.07) | 1907.5 (153.91) | 2411.8 (218.29) | 2349.3 (210.77)

8. Secondary Outcome: Geometric Mean of the Maximum Observed Plasma Concentration (Cmax) for Pramlintide at Weeks 4 and 24 - Evaluable Population Receiving Pramlintide
Description: Assessment of Cmax was over a period of 2 hours following pramlintide administration at Weeks 4 and 24. Cmax was measured as picograms/milliliter (pg/mL).
Time Frame: Week 4 and Week 24
Population: Evaluable population: participants received at least one dose of randomized treatment, had adequate exposure to treatment and complied with the protocol as assessed prior to database lock and unblinding. Number (n) analyzed at Week 4 n=46,40,41,40,40,33 in each arm, respectively; Week 24 n=48,38, 44,40,35,36 in each arm, respectively.
Measure: Geometric Mean (Standard Error); unit: pg/mL
Arm/Group | Pramlintide 360 mcg + Placebo-M | Pramlintide 180 mcg + Metreleptin 2.5 mg | Pramlintide 180 mcg + Metreleptin 5.0 mg | Pramlintide 360 mcg + Metreleptin 1.25 mg | Pramlintide 360 mcg + Metreleptin 2.5 mg | Pramlintide 360 mcg + Metreleptin 5.0 mg
Number analyzed (Participants) | 48 | 40 | 44 | 40 | 40 | 36
pg/mL
  Week 4 Cmax | 1759.0 (168.40) | 876.7 (77.37) | 897.3 (51.16) | 1783.8 (144.34) | 1851.3 (118.87) | 2096.4 (149.65)
  Week 24 Cmax | 1985.8 (118.31) | 1048.1 (76.86) | 925.5 (64.16) | 1573.5 (100.69) | 2032.0 (152.70) | 1972.2 (159.33)

9. Secondary Outcome: Least Squares (LS) Mean Absolute Change From Baseline to Week 28 in Percent of Body Fat - Evaluable Population
Description: Parameters of body composition were measured with a Dual Energy X-ray absorptiometry (DEXA) scan and reported as a percent (%). Data from the first valid DEXA scan obtained no later than 7 days after the first randomized dose was considered as valid baseline values; data from the last valid DEXA scan obtained no later than 10 days after last clinical visit or no later than 14 days after last dose of randomized study medication was considered as valid study termination values. Absolute change from baseline was defined as percent body fat at Week 28 - percent body fat at baseline.
Time Frame: Baseline to Week 28
Population: Evaluable population includes participants received at least one dose of randomized treatment, had adequate exposure to treatment, and complied with the protocol as assessed prior to database lock and unblinding. Number analyzed (n) were of evaluable participants with valid DEXA scan at Week 28.
Measure: Least Squares Mean (Standard Error); unit: percentage of body fat
Arm/Group | Placebo | Pramlintide 360 mcg | Metreleptin 5.0 mg | Pramlintide 180 mcg + Metreleptin 2.5 mg | Pramlintide 180 mcg + Metreleptin 5.0 mg | Pramlintide 360 mcg + Metreleptin 1.25 mg | Pramlintide 360 mcg + Metreleptin 2.5 mg | Pramlintide 360 mcg + Metreleptin 5.0 mg
Number analyzed (Participants) | 36 | 51 | 38 | 40 | 42 | 39 | 40 | 35
percentage of body fat | -0.95 (0.501) | -1.77 (0.421) | -1.94 (0.492) | -2.32 (0.480) | -2.21 (0.475) | -2.21 (0.497) | -1.56 (0.482) | -2.46 (0.515)
Statistical Analysis 1: Comparison: Placebo vs Pramlintide 180 mcg + Metreleptin 2.5 mg; Based on a general linear model general linear model that includes baseline value and factors for treatment group, sex, baseline BMI category (<35 kg/m2, 35 to <40 kg/m2, ≥40 kg/m2); Test type: Superiority or Other; p = 0.0464, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo vs Pramlintide 180 mcg + Metreleptin 5.0 mg; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.0647, t-test, 2 sided
Statistical Analysis 3: Comparison: Placebo vs Pramlintide 360 mcg + Metreleptin 1.25 mg; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.0690, t-test, 2 sided
Statistical Analysis 4: Comparison: Placebo vs Pramlintide 360 mcg + Metreleptin 2.5 mg; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.3717, t-test, 2 sided
Statistical Analysis 5: Comparison: Placebo vs Pramlintide 360 mcg + Metreleptin 5.0 mg; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.0327, t-test, 2 sided

10. Secondary Outcome: LS Mean Absolute Change From Baseline to Week 28 in Total Body Fat Mass (k) - Evaluable Population
Description: Parameters of body composition were measured with a Dual Energy X-ray absorptiometry (DEXA) scan. Data from the first valid DEXA scan obtained no later than 7 days after the first randomized dose was considered as valid baseline values; data from the last valid DEXA scan obtained no later than 10 days after last clinical visit or no later than 14 days after last dose of randomized study medication was considered as valid study termination values. Body fat mass was measured in kilogram (k).
Time Frame: Baseline to Week 28
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo | Pramlintide 360 mcg | Metreleptin 5.0 mg | Pramlintide 180 mcg + Metreleptin 2.5 mg | Pramlintide 180 mcg + Metreleptin 5.0 mg | Pramlintide 360 mcg + Metreleptin 1.25 mg | Pramlintide 360 mcg + Metreleptin 2.5 mg | Pramlintide 360 mcg + Metreleptin 5.0 mg
Number analyzed (Participants) | 36 | 51 | 38 | 40 | 42 | 39 | 40 | 35
kg | -1.96 (0.0779) | -4.28 (0.661) | -4.57 (0.763) | -4.98 (0.746) | -4.97 (0.734) | -5.03 (0.755) | -4.35 (0.748) | -5.51 (0.792)
Statistical Analysis 1: Comparison: Placebo vs Pramlintide 180 mcg + Metreleptin 2.5 mg; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.0049, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo vs Pramlintide 180 mcg + Metreleptin 5.0 mg; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.0047, t-test, 2 sided
Statistical Analysis 3: Comparison: Placebo vs Pramlintide 360 mcg + Metreleptin 1.25 mg; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.0046, t-test, 2 sided
Statistical Analysis 4: Comparison: Placebo vs Pramlintide 360 mcg + Metreleptin 2.5 mg; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.0257, t-test, 2 sided
Statistical Analysis 5: Comparison: Placebo vs Pramlintide 360 mcg + Metreleptin 5.0 mg; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.0014, t-test, 2 sided

11. Secondary Outcome: LS Mean Absolute Change From Baseline to Week 28 in Fat-free Mass (kg) - Evaluable Population
Description: Parameters of body composition were measured with a Dual Energy X-ray Absorptiometry (DEXA) scan. Data from the first valid DEXA scan obtained no later than 7 days after the first randomized dose was considered as valid baseline values; data from the last valid DEXA scan obtained no later than 10 days after last clinical visit or no later than 14 days after last dose of randomized study medication was considered as valid study termination values. Fat-free mass were measured in kilogram (k).
Time Frame: Baseline to Week 28
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo | Pramlintide 360 mcg | Metreleptin 5.0 mg | Pramlintide 180 mcg + Metreleptin 2.5 mg | Pramlintide 180 mcg + Metreleptin 5.0 mg | Pramlintide 360 mcg + Metreleptin 1.25 mg | Pramlintide 360 mcg + Metreleptin 2.5 mg | Pramlintide 360 mcg + Metreleptin 5.0 mg
Number analyzed (Participants) | 36 | 51 | 38 | 40 | 42 | 39 | 40 | 35
kg | -0.69 (0.393) | -1.62 (0.337) | -1.80 (0.389) | -1.90 (0.377) | -1.99 (0.373) | -2.02 (0.391) | -2.11 (0.380) | -2.29 (0.399)
Statistical Analysis 1: Comparison: Placebo vs Pramlintide 180 mcg + Metreleptin 2.5 mg; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.0222, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo vs Pramlintide 180 mcg + Metreleptin 5.0 mg; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.0128, t-test, 2 sided
Statistical Analysis 3: Comparison: Placebo vs Pramlintide 360 mcg + Metreleptin 1.25 mg; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.0122, t-test, 2 sided
Statistical Analysis 4: Comparison: Placebo vs Pramlintide 360 mcg + Metreleptin 2.5 mg; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.0073, t-test, 2 sided
Statistical Analysis 5: Comparison: Placebo vs Pramlintide 360 mcg + Metreleptin 5.0 mg; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.0034, t-test, 2 sided

12. Secondary Outcome: LS Mean Absolute Change From Baseline to Week 28 in Fasting Plasma Glucose, Total Cholesterol (TC), Triglycerides, Low Density Lipoprotein (LDL) Cholesterol, High Density Lipoprotein (HDL) Cholesterol - Evaluable Population
Description: Baseline refers to Visit 5 (Day 1). If Day 1 value is missing or after the first dose date of randomized study medication, the last available value on or prior to Day 1 is used. Fasting samples were obtained at baseline, Weeks 4, 12, and 28. All parameters were measured in milligrams per deciliter (mg/dL).
Time Frame: Baseline to Week 28
Population: Evaluable population: received at least one dose of randomized treatment, had adequate exposure to treatment, complied with the protocol as assessed prior to database lock and unblinding. Number analyzed (n) presented above for TC, LDL and HDL cholesterol. Glucose n= 43, 50, 41, 46, 45, 43,44,36; Triglycerides n= 44,50,41,46,45,44,44.38.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Pramlintide 360 mcg | Metreleptin 5.0 mg | Pramlintide 180 mcg + Metreleptin 2.5 mg | Pramlintide 180 mcg + Metreleptin 5.0 mg | Pramlintide 360 mcg + Metreleptin 1.25 mg | Pramlintide 360 mcg + Metreleptin 2.5 mg | Pramlintide 360 mcg + Metreleptin 5.0 mg
Number analyzed (Participants) | 44 | 50 | 39 | 46 | 45 | 44 | 44 | 37
mg/dL
  Fasting Plasma Glucose | -1.3 (1.35) | -1.8 (1.25) | -1.8 (1.39) | -2.5 (1.32) | -1.2 (1.34) | -1.0 (1.36) | -1.7 (1.35) | -1.3 (1.47)
  Total Cholesterol | 4.3 (3.57) | -7.1 (3.35) | -3.7 (3.82) | -2.1 (3.54) | -2.5 (3.60) | -0.6 (3.60) | -4.0 (3.61) | -1.3 (3.88)
  Triglycerides | -0.1 (8.25) | -8.6 (7.73) | -13.0 (8.66) | -1.4 (8.17) | -10.9 (8.29) | 11.1 (8.34) | -9.2 (8.35) | 0.9 (8.86)
  LDL Cholesterol | 4.3 (2.82) | -3.5 (2.65) | -2.3 (3.02) | -3.7 (2.80) | -0.0 (2.85) | -2.7 (2.85) | -3.7 (2.86) | -1.2 (3.08)
  HDL Cholesterol | 1.5 (0.96) | 0.6 (0.90) | 2.6 (1.03) | 0.7 (0.95) | 1.0 (0.96) | 2.9 (0.97) | 0.97 (0.97) | 1.05 (1.05)

13. Secondary Outcome: Mean Absolute Change From Baseline to Week 28 for Insulin - Evaluable Population
Description: Baseline refers to Visit 5 (Day 1). If Day 1 value is missing or after the first dose date of randomized study medication, the last available value on or prior to Day 1 is used. Fasting samples were obtained at baseline, Weeks 4, 12, and 28. Parameter was measured micro international units per milliliter. (µIU/mL).
Time Frame: Baseline to Week 28
Population: Evaluable population includes participants received at least one dose of randomized treatment, had adequate exposure to treatment, and complied with the protocol as assessed prior to database lock and unblinding.
Measure: Least Squares Mean (Standard Error); unit: µIU/mL
Arm/Group | Placebo | Pramlintide 360 mcg | Metreleptin 5.0 mg | Pramlintide 180 mcg + Metreleptin 2.5 mg | Pramlintide 180 mcg + Metreleptin 5.0 mg | Pramlintide 360 mcg + Metreleptin 1.25 mg | Pramlintide 360 mcg + Metreleptin 2.5 mg | Pramlintide 360 mcg + Metreleptin 5.0 mg
Number analyzed (Participants) | 42 | 49 | 40 | 44 | 45 | 43 | 43 | 36
µIU/mL | 1.1 (1.01) | -0.4 (0.94) | -1.6 (1.0) | -1.0 (1.00) | -2.5 (0.99) | -1.4 (1.00) | -0.8 (1.01) | -0.5 (1.08)

14. Secondary Outcome: Mean Absolute Change From Screening to Week 24 in Impact of Weight on Quality of Life Questionnaire-lite Version (IWQOL-Lite) Total Score - Evaluable Population
Description: Subjective effects of weight loss were measured using the IWQOL-Lite questionnaire, a 31-item patient reported outcome (PRO) instrument used to assess the effect of weight on physical function, self-esteem, sexual life, public distress, and work. Individual items have a range of 1 to 5 with 5=always true and 1= never true. The total score for the IWQOL-Lite instrument is measured on a scale from 0 (worst) to 100 (best). Higher scores indicate improvement. Values were obtained for this questionnaire on Visit 3 in the screening period.
Time Frame: Screening to Week 24
Population: Evaluable population includes participants received at least one dose of randomized treatment, had adequate exposure to treatment, and complied with the protocol as assessed prior to database lock and unblinding. Missing item responses may be imputed for each subject as appropriate before summarization.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pramlintide 360 mcg | Metreleptin 5.0 mg | Pramlintide 180 mcg + Metreleptin 2.5 mg | Pramlintide 180 mcg + Metreleptin 5.0 mg | Pramlintide 360 mcg + Metreleptin 1.25 mg | Pramlintide 360 mcg + Metreleptin 2.5 mg | Pramlintide 360 mcg + Metreleptin 5.0 mg
Number analyzed (Participants) | 46 | 51 | 41 | 47 | 46 | 44 | 45 | 35
units on a scale | 10.52 (12.480) | 10.31 (11.629) | 11.09 (13.503) | 10.14 (10.957) | 16.15 (15.193) | 13.84 (11.535) | 13.44 (11.175) | 11.68 (10.271)

15. Secondary Outcome: Mean Absolute Change From Screening to Week 24 in Binge Eating Scale (BES) Total Score - Evaluable Population
Description: The Binge Eating Scale (BES) is a 16-item questionnaire that assesses the behavioral and cognitive correlates of binge eating, including participants' perceived self-control over eating behavior using a range of 1 to 4 with 1=positive perceptions and 4= negative perceptions. The minimum and maximum score for the BES instrument is 0 and 55, respectively. The higher the score the worse the outcome. Values were obtained for this questionnaire on Visit 3 in the screening period.
Time Frame: Screening to Week 24
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pramlintide 360 mcg | Metreleptin 5.0 mg | Pramlintide 180 mcg + Metreleptin 2.5 mg | Pramlintide 180 mcg + Metreleptin 5.0 mg | Pramlintide 360 mcg + Metreleptin 1.25 mg | Pramlintide 360 mcg + Metreleptin 2.5 mg | Pramlintide 360 mcg + Metreleptin 5.0 mg
Number analyzed (Participants) | 46 | 49 | 41 | 47 | 46 | 43 | 45 | 36
units on a scale | -3.0 (6.31) | -3.4 (6.96) | -4.0 (6.21) | -4.4 (6.45) | -6.6 (8.28) | -3.5 (5.87) | -5.9 (7.44) | -5.2 (6.17)

16. Secondary Outcome: Mean Absolute Change From Screening to Week 24 in Susceptibility to Eating Questionnaire (SEQ) Item Scores - Evaluable Population
Description: The eating questionnaire is an exploratory measure of appetite, satiety, and perceived control over portion size using 10 VAS items with each response measured on a 100 mm visual analogue scale (ranges vary from Never to Very Often; Not at All Difficult to Extremely Difficult; Not at all Strong to Very Strong). Lower scores indicate improvement. The Eating Questionnaire instructed participants to rate their responses to these items over the past 7 days. Values were obtained for this questionnaire on Visit 3 in the screening period.
Time Frame: Screening to Week 24
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pramlintide 360 mcg | Metreleptin 5.0 mg | Pramlintide 180 mcg + Metreleptin 2.5 mg | Pramlintide 180 mcg + Metreleptin 5.0 mg | Pramlintide 360 mcg + Metreleptin 1.25 mg | Pramlintide 360 mcg + Metreleptin 2.5 mg | Pramlintide 360 mcg + Metreleptin 5.0 mg
Number analyzed (Participants) | 46 | 51 | 41 | 47 | 45 | 44 | 45 | 36
units on a scale
  Frequency of Food Cravings | -9.0 (25.85) | -6.6 (27.17) | -4.0 (24.28) | -14.1 (24.55) | -19.8 (31.06) | -15.7 (21.76) | -18.5 (27.69) | -13.5 (29.56)
  Strength of Food Cravings | -5.1 (27.60) | -6.1 (26.86) | -1.1 (24.97) | -13.9 (25.45) | -13.8 (28.02) | -12.9 (19.19) | -19.6 (25.66) | -15.2 (32.56)
  Difficult to Control Eating | -8.1 (27.45) | -15.2 (26.37) | -9.5 (27.44) | -19.7 (23.00) | -27.3 (27.02) | -18.3 (19.46) | -26.3 (28.89) | -18.0 (35.40)
  Difficult to Resist Food Cravings | -11.4 (30.32) | -11.1 (24.52) | 9.6 (25.02) | -19.5 (26.28) | -21.8 (28.65) | -19.0 (26.49) | -28.0 (29.90) | -18.2 (29.80)
  Eating in Response to Food Cravings | -11.1 (28.41) | -12.2 (25.14) | -12.6 (27.34) | -15.4 (22.17) | -22.2 (32.94) | -18.5 (24.95) | -22.9 (27.85) | -15.9 (27.04)
  Difficult to Control Portion Sizes | -10.8 (23.37) | -16.9 (29.58) | -27.6 (30.70) | -19.6 (21.19) | -25.2 (28.00) | -20.8 (21.18) | -24.0 (26.91) | -27.6 (34.18)
  How Hungry | -0.1 (20.59) | -9.7 (22.92) | -17.5 (23.18) | -16.4 (24.00) | -17.0 (24.09) | -17.5 (22.53) | -19.2 (24.64) | -19.9 (31.32)
  How Full After Meals | -5.8 (25.37) | 0.5 (25.05) | -7.6 (19.94) | -3.8 (26.19) | -8.8 (31.83) | -6.5 (26.46) | -4.2 (27.71) | 1.1 (23.42)
  Thoughts of Food | -2.7 (21.70) | -10.7 (25.84) | -10.6 (30.04) | -9.4 (22.33) | -16.7 (27.75) | -12.0 (20.98) | -20.0 (27.90) | -5.6 (30.73)
  How Pleasant Meals | -6.1 (19.72) | -2.3 (24.55) | -2.1 (21.00) | 1.2 (27.11) | -1.2 (25.96) | 3.7 (24.87) | 5.3 (22.41) | -2.1 (28.08)

17. Secondary Outcome: Mean Absolute Change From Screening to Week 24 in Hospital Anxiety and Depression Scale (HADS) Total Scores - Evaluable Population
Description: The HADS is a questionnaire that uses 14 items to assess both anxiety and depression over the past week. The odd numbered items constitute the anxiety subscale, and the even numbered items constitute the depression subscale. The individual response scores for each subscale component are added together to obtain the individual subscale scores. The minimum and maximum score for each subscale is 0 and 21, respectively. The higher the score, the worse the outcome. Values were obtained for this questionnaire on Visit 3 in the screening period
Time Frame: Screening to Week 24
Population: as for outcome 14
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Pramlintide 360 mcg | Metreleptin 5.0 mg | Pramlintide 180 mcg + Metreleptin 2.5 mg | Pramlintide 180 mcg + Metreleptin 5.0 mg | Pramlintide 360 mcg + Metreleptin 1.25 mg | Pramlintide 360 mcg + Metreleptin 2.5 mg | Pramlintide 360 mcg + Metreleptin 5.0 mg
Number analyzed (Participants) | 46 | 51 | 41 | 47 | 46 | 44 | 45 | 36
units on a scale
  Anxiety Total Scores | 0.02 (0.475) | 0.08 (0.274) | -0.56 (0.342) | -0.11 (0.431) | -0.43 (0.373) | -0.59 (0.370) | -0.58 (0.429) | 0.06 (0.465)
  Depression Total Scores | -0.85 (0.435) | -0.76 (0.357) | -0.98 (0.394) | -0.66 (0.332) | -1.37 (0.387) | -1.23 (0.416) | -1.02 (0.294) | 0.00 (0.481)

18. Secondary Outcome: Mean Absolute Change From Screening to Week 24 in Summary Scores for Profile of Mood States - Brief (POMS-B) - Evaluable Population
Description: The POMS is a mood scale consisting of 65 mood adjectives that assess participants' mood over the past seven days. The POMS-B is an authorized, 30-item brief version of the POMS consisting of five items for each of the six POMS factors. The mood adjectives load onto 6 mood factors, which are as follows: Tension-Anxiety, Depression-Dejection, Anger-Hostility, Vigor-Activity, Fatigue-Inertia, and Confusion-Bewilderment. Scores range from 0= Not at All to 4=Extremely. The factor scores are added to obtain the total mood disturbance score. A lower total mood disturbance score indicates improvement. Values were obtained for this questionnaire on Visit 3 in the screening period.
Time Frame: Screening to Week 24
Population: as for outcome 14
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Pramlintide 360 mcg | Metreleptin 5.0 mg | Pramlintide 180 mcg + Metreleptin 2.5 mg | Pramlintide 180 mcg + Metreleptin 5.0 mg | Pramlintide 360 mcg + Metreleptin 1.25 mg | Pramlintide 360 mcg + Metreleptin 2.5 mg | Pramlintide 360 mcg + Metreleptin 5.0 mg
Number analyzed (Participants) | 46 | 51 | 41 | 47 | 46 | 43 | 45 | 35
units on a scale
  Tension - Anxiety | 0.35 (0.518) | 0.39 (0.308) | -0.17 (0.389) | 0.87 (0.518) | -0.30 (0.408) | -0.21 (0.358) | 0.00 (0.423) | 0.66 (0.583)
  Depression - Dejection | 0.41 (0.628) | 0.27 (0.489) | 0.44 (0.466) | 0.64 (0.410) | 0.26 (0.464) | 0.37 (0.381) | -0.29 (0.348) | 0.23 (0.666)
  Anger - Hostility | 0.04 (0.577) | 0.16 (0.418) | -0.22 (0.468) | 0.53 (0.489) | -0.30 (0.409) | -0.05 (0.410) | -0.18 (0.476) | 0.71 (0.515)
  Vigor - Activity | 1.11 (0.534) | 0.27 (0.681) | 0.78 (0.670) | 1.04 (0.603) | 1.20 (0.632) | 0.95 (0.773) | 1.13 (0.641) | 1.29 (0.787)
  Fatigue - Inertia | -1.22 (0.852) | -0.53 (0.709) | -1.10 (0.688) | 0.02 (0.660) | -0.30 (0.676) | -1.49 (0.626) | -0.82 (0.667) | 0.09 (0.779)
  Confusion - Bewilderment | 0.43 (0.471) | 0.51 (0.334) | 0.17 (0.296) | 0.40 (0.387) | 0.20 (0.400) | 0.05 (0.286) | 0.02 (0.280) | 0.00 (0.393)

19. Secondary Outcome: Mean Absolute Change From Screening to Week 24 in Minutes to Fall Asleep, Hours of Sleep and The Pittsburgh Sleep Quality Index (PSQI) Global Score - Evaluable Population
Description: The Pittsburgh Sleep Quality Index (PSQI) is a questionnaire which assesses sleep quality and sleep disturbances over a period of 1 month. The PSQI provides ratings on seven domains of sleep (subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction). The sum of the individual domains yields a global sleep quality score with a range of 0-21. A PSQI score >5 is indicative of poor sleep, which is characterized by severe difficulties in at least two domains, or moderate difficulties in three or more domains. Values were obtained for this questionnaire on Visit 3 in the screening period.
Time Frame: Screening to Week 24
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pramlintide 360 mcg | Metreleptin 5.0 mg | Pramlintide 180 mcg + Metreleptin 2.5 mg | Pramlintide 180 mcg + Metreleptin 5.0 mg | Pramlintide 360 mcg + Metreleptin 1.25 mg | Pramlintide 360 mcg + Metreleptin 2.5 mg | Pramlintide 360 mcg + Metreleptin 5.0 mg
Number analyzed (Participants) | 46 | 51 | 41 | 47 | 46 | 45 | 45 | 38
units on a scale
  Minutes to Fall Asleep | -0.5 (11.17) | 1.3 (17.83) | -2.1 (14.81) | -4.3 (15.09) | -4.6 (12.00) | -4.3 (19.50) | -1.0 (14.74) | 2.7 (16.04)
  Hours Asleep | 0.1 (0.80) | 0.1 (0.91) | -0.1 (0.76) | 0.2 (1.09) | 0.1 (1.15) | 0.2 (1.01) | 0.2 (1.18) | -0.4 (1.06)
  PSQI Global Score | -0.9 (2.18) | -0.3 (2.46) | -0.3 (2.81) | -0.8 (2.43) | -0.9 (2.92) | -1.0 (2.57) | -1.0 (2.44) | -0.1 (2.64)

20. Secondary Outcome: Mean Absolute Change From Screening to Week 24 in the Epworth Sleepiness Scale (ESS) Total Score - Evaluable Population
Description: The Epworth Sleepiness Scale (ESS) is an eight-item questionnaire that assesses sleep propensity in daily situations of increasing sleepiness on a four-point scale with 0=would never doze and 3=high chance of dozing. Lower scores indicate improvement. Values were obtained for this questionnaire on Visit 3 in the screening period
Time Frame: Screening to Week 24
Population: as for outcome 14
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Pramlintide 360 mcg | Metreleptin 5.0 mg | Pramlintide 180 mcg + Metreleptin 2.5 mg | Pramlintide 180 mcg + Metreleptin 5.0 mg | Pramlintide 360 mcg + Metreleptin 1.25 mg | Pramlintide 360 mcg + Metreleptin 2.5 mg | Pramlintide 360 mcg + Metreleptin 5.0 mg
Number analyzed (Participants) | 45 | 51 | 41 | 47 | 46 | 44 | 45 | 36
units on a scale | -0.69 (0.552) | -0.63 (0.450) | 0.12 (0.621) | -1.32 (0.319) | -1.80 (0.426) | -1.05 (0.662) | -1.80 (0.448) | -0.42 (0.522)

21. Secondary Outcome: Number of Hematology and Urinalysis Laboratory Values of Potential Clinical Importance Observed From Screening to Week 28 - Intent to Treat Population
Description: Criteria for laboratory values of potential clinical importance for obese and overweight (BMI >= 25 kg/m^2) participants: Platelets high (H) >500,000/µL; low (L) <75,000/µL. Hematocrit males <36%, females <30%. Hemoglobin males <12 g/dL, females <10 g/dL. White blood cell count (WBC) H >18,000/µL; L <1,500/µL. Urine protein H >= 3+ or >= 500 mg/dL. Urine glucose H >= 3+ or >= 500 mg/dL. Urine ketones >= 3+ or Large. Values obtained at Screening, Day -7, Day 1, Weeks 1, 2, 4, 8, 12, 16, 20, 24, 28. Numbers of values are cumulative across the study.
Time Frame: Screening to Week 28
Population: Intent to treat population included all randomized participants who received at least one injection of study medication.
Measure: Number; unit: Number of Laboratory Values
Arm/Group | Placebo | Pramlintide 360 mcg | Metreleptin 5.0 mg | Pramlintide 180 mcg + Metreleptin 2.5 mg | Pramlintide 180 mcg + Metreleptin 5.0 mg | Pramlintide 360 mcg + Metreleptin 1.25 mg | Pramlintide 360 mcg + Metreleptin 2.5 mg | Pramlintide 360 mcg + Metreleptin 5.0 mg
Number analyzed (Participants) | 75 | 77 | 72 | 75 | 78 | 78 | 78 | 75
Number of Laboratory Values
  Hematocrit | 4 | 0 | 0 | 0 | 0 | 1 | 4 | 3
  Hemoglobin | 7 | 0 | 0 | 0 | 0 | 5 | 7 | 4
  Platelet Count | 0 | 0 | 1 | 1 | 0 | 0 | 10 | 0
  White Blood Cell Count | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urine Glucose | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Urine Ketones | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Urine protein | 1 | 2 | 0 | 2 | 3 | 4 | 2 | 1

22. Secondary Outcome: Number of Chemistry Laboratory Values of Potential Clinical Importance Observed From Screening to Week 28 - Intent to Treat Population
Description: Obtained at: Screening, Days -7, 1, Weeks 1, 2, 4, 8, 12, 16, 20, 24, 28. Numbers of laboratory values are cumulative across the study. Criteria for values of potential clinical importance for obese and overweight (BMI>=25 kg/m^2) participants: Total bilirubin High (H) > 2 mg/dL; Plasma/serum glucose fasting or non-fasting H > 200 mg/dL, low (L) < 60 mg/dL; Albumin L <2.5 g/dL; Creatine kinase H > 3*Upper limit of Normal (ULN); Sodium L <130 milliequivalents per liter (mEq/L), H > 150 mEq/L; potassium L<3.0 mEq/L, H> 5.5 mEq/L;bicarbonate L<18 mEq/L, H>35 mEq/L;calcium L <8mg/dL, H> 11 mg/dL; triglycerides H> 500 mg/dL; Cholesterol L < 100 mg/dL, H > 350 mg/dL; Alkaline phosphatase H > 3*ULN; Gamma-glutamyltransferase H>3*ULN; creatinine males > 1.6 mg/dL, females > 1.4 mg/dL; alanine aminotransferase H > 3*ULN; aspartate aminotransferase H > 3*ULN; urea nitrogen H > 45 mg/dL; uric acid males > 10.0 mg/dL, females > 8.0 mg/dL; Phosphorus L < 1.0 mg/dL H > 6.0 mg/dL.
Time Frame: Screening to Week 28
Population: Intent to treat population included all randomized participants who received at least one injection of study medication.
Measure: Number; unit: Number of Laboratory Values
Arm/Group | Placebo | Pramlintide 360 mcg | Metreleptin 5.0 mg | Pramlintide 180 mcg + Metreleptin 2.5 mg | Pramlintide 180 mcg + Metreleptin 5.0 mg | Pramlintide 360 mcg + Metreleptin 1.25 mg | Pramlintide 360 mcg + Metreleptin 2.5 mg | Pramlintide 360 mcg + Metreleptin 5.0 mg
Number analyzed (Participants) | 75 | 77 | 72 | 75 | 78 | 78 | 78 | 75
Number of Laboratory Values
  alanine aminotransferase | 0 | 8 | 1 | 0 | 0 | 0 | 0 | 3
  aspartate aminotransferase | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 2
  Bicarbonate | 0 | 5 | 1 | 5 | 1 | 0 | 0 | 1
  Gamma-glutamyltransferase | 17 | 3 | 5 | 1 | 13 | 0 | 0 | 6
  Creatine kinase | 18 | 4 | 4 | 9 | 8 | 4 | 2 | 2
  Calcium | 2 | 2 | 2 | 7 | 1 | 0 | 13 | 0
  Potassium | 0 | 1 | 0 | 1 | 2 | 1 | 2 | 6
  Sodium | 2 | 4 | 2 | 4 | 2 | 0 | 3 | 0
  Creatinine | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 3
  Total Bilirubin | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Uric Acid | 4 | 10 | 5 | 11 | 19 | 21 | 9 | 25
  Alkaline Phosphatase | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Blood urea nitrogen | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

23. Secondary Outcome: Mean Change in Systolic and Diastolic Blood Pressure From Baseline to Week 28 - Intent to Treat Population
Description: Baseline refers to Day 1. If Day 1 value was missing or after the first dose date of randomized study medication, the last available value on or prior to Day 1 was used. Blood pressure was taken while the participant was sitting and was measured in millimeters of mercury (mm Hg). Values obtained at Screening, Day -7, Day 1, Weeks 1, 2, 4, 8, 12, 16, 20, 24, 28
Time Frame: Baseline to Week 28
Population: Intent to treat population included all randomized participants who received at least one injection of study medication.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Pramlintide 360 mcg | Metreleptin 5.0 mg | Pramlintide 180 mcg + Metreleptin 2.5 mg | Pramlintide 180 mcg + Metreleptin 5.0 mg | Pramlintide 360 mcg + Metreleptin 1.25 mg | Pramlintide 360 mcg + Metreleptin 2.5 mg | Pramlintide 360 mcg + Metreleptin 5.0 mg
Number analyzed (Participants) | 75 | 77 | 72 | 75 | 78 | 78 | 78 | 75
mm Hg
  Systolic Blood Pressure | 2.4 (10.65) | -0.9 (11.9) | -3.4 (12.54) | -3.2 (10.84) | 0.4 (11.84) | -2.0 (12.47) | -1.2 (10.78) | -1.5 (12.54)
  Diastolic Blood Pressure | 1.2 (7.31) | -1.7 (6.83) | -2.6 (7.21) | -0.4 (8.07) | -1.0 (6.99) | -1.3 (7.96) | -1.8 (6.77) | -0.1 (9.93)

24. Secondary Outcome: Mean Change in Heart Rate From Baseline to Week 28 - Intent to Treat Population
Description: Baseline refers to Day 1. If Day 1 value was missing or after the first dose date of randomized study medication, the last available value on or prior to Day 1 was used. Heart rate was measured while the participant was sitting and was measured in beats per minute (bpm). Values obtained at Screening, Day -7, Day 1, Weeks 1, 2, 4, 8, 12, 16, 20, 24, 28.
Time Frame: Baseline to Week 28
Population: Intent to treat population included all randomized participants who received at least one injection of study medication.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Placebo | Pramlintide 360 mcg | Metreleptin 5.0 mg | Pramlintide 180 mcg + Metreleptin 2.5 mg | Pramlintide 180 mcg + Metreleptin 5.0 mg | Pramlintide 360 mcg + Metreleptin 1.25 mg | Pramlintide 360 mcg + Metreleptin 2.5 mg | Pramlintide 360 mcg + Metreleptin 5.0 mg
Number analyzed (Participants) | 74 | 77 | 72 | 75 | 78 | 78 | 78 | 75
bpm | 1.6 (9.29) | -1.3 (7.70) | -2.6 (6.66) | -1.4 (8.40) | -2.1 (7.38) | -0.5 (9.34) | -2.4 (7.54) | -0.1 (10.80)

25. Secondary Outcome: Number of Participants With Treatment-emergent Positive Anti-leptin Antibody Titers at Week 28 - Intent to Treat Population
Description: Baseline refers to Day 1. If Day 1 value was missing or after the first dose date of randomized study medication, the last available value on or prior to Day 1 was used. Serum titer determinations for antibodies to metreleptin were made using a validated electrochemical luminescence (ECLA) bridging assay. Antibody titers were assessed according to the following dilutions: 0, 5, 25, 125, 625, 3125, 15625, and 78125. Participants were considered to have a positive titer to treatment-emergent antibodies to metreleptin at a given visit if they had a titer >=5 following a negative or missing titer at baseline or if they had a titer that had increased by at least 2 dilutions from a detectable level at baseline.
Time Frame: Baseline to Week 28
Population: Intent to treat population included all randomized participants who received at least one injection of study medication.
Measure: Number; unit: participants
Arm/Group | Metreleptin 5.0 mg | Pramlintide 180 mcg + Metreleptin 2.5 mg | Pramlintide 180 mcg + Metreleptin 5.0 mg | Pramlintide 360 mcg + Metreleptin 1.25 mg | Pramlintide 360 mcg + Metreleptin 2.5 mg | Pramlintide 360 mcg + Metreleptin 5.0 mg
Number analyzed (Participants) | 45 | 49 | 50 | 44 | 50 | 43
participants | 43 | 49 | 48 | 42 | 50 | 42

26. Secondary Outcome: Mean Change From Screening to Week 28 in Electrocardiogram Parameters - Intent to Treat Population
Description: A 12-Lead electrocardiogram (ECG) was obtained at Screening, Day 1, Weeks 1, 12, 28 (study termination). The PR interval, which is time from beginning of the P wave to the beginning of the QRS complex (Note: QRS complex is a name for the combination of 3 of the graphical deflections seen in an ECG); QRS interval (time from the beginning to the end of the QRS complex); QT interval (measure between Q wave and T wave in the heart's electrical cycle); and QT interval corrected for heart rate using Fridericia's formula (QTcF) were measured in milliseconds (msec).
Time Frame: Screening to Week 28 (or study termination)
Population: Intent to treat population included all randomized participants who received at least one injection of study medication.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Placebo | Pramlintide 360 mcg | Metreleptin 5.0 mg | Pramlintide 180 mcg + Metreleptin 2.5 mg | Pramlintide 180 mcg + Metreleptin 5.0 mg | Pramlintide 360 mcg + Metreleptin 1.25 mg | Pramlintide 360 mcg + Metreleptin 2.5 mg | Pramlintide 360 mcg + Metreleptin 5.0 mg
Number analyzed (Participants) | 46 | 54 | 41 | 49 | 47 | 44 | 47 | 39
msec
  PR Interval | 1.1 (12.73) | -0.1 (12.23) | 0.3 (10.37) | 0.1 (13.74) | 16.8 (97.51) | 4.4 (17.89) | 0.4 (11.86) | -1.6 (14.27)
  QRS Interval | -0.3 (5.20) | -1.4 (8.76) | 1.0 (4.66) | -0.5 (6.26) | -1.8 (5.62) | -0.2 (4.12) | 0.3 (4.78) | -0.4 (5.33)
  QT Interval | 0.4 (28.72) | 9.9 (21.80) | 16.2 (28.64) | 7.0 (19.33) | 8.9 (20.53) | 4.4 (24.97) | 15.0 (21.56) | 6.3 (28.03)
  QTcF | -0.3 (21.75) | 4.0 (15.58) | 8.2 (21.39) | -1.2 (16.02) | -0.8 (15.13) | 0.3 (15.40) | 1.3 (12.34) | -2.3 (22.00)

27. Secondary Outcome: Mean Change From Screening to Week 28 in the Electrocardiogram Parameter of Heart Rate - Intent to Treat Population
Description: A 12-Lead electrocardiogram (ECG) was obtained at Screening (visit 2), Day 1, Weeks 1, 12, 28 (study termination). Heart Rate was measured in beats per min (bpm).
Time Frame: Screening to Week 28 (or early termination)
Population: Intent to treat population included all randomized participants who received at least one injection of study medication.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Placebo | Pramlintide 360 mcg | Metreleptin 5.0 mg | Pramlintide 180 mcg + Metreleptin 2.5 mg | Pramlintide 180 mcg + Metreleptin 5.0 mg | Pramlintide 360 mcg + Metreleptin 1.25 mg | Pramlintide 360 mcg + Metreleptin 2.5 mg | Pramlintide 360 mcg + Metreleptin 5.0 mg
Number analyzed (Participants) | 46 | 54 | 41 | 49 | 47 | 44 | 47 | 39
bpm | 0.3 (13.96) | -2.8 (8.45) | -4.1 (8.18) | -4.7 (10.12) | -4.9 (9.42) | -1.9 (9.73) | -6.6 (8.41) | -3.4 (9.69)

ADVERSE EVENTS:
Time Frame: From enrollment to Study Termination (Week 28). Clinically significant events that continued beyond termination were followed until diagnosis/resolution occurred. Serious adverse events were followed 30 days post last dose of study medication.
Description: All participants enrolled were treated with Placebo for 1 week and then randomized into a treatment group. Enrolled = 636 (commenced placebo for 1 week); Enrolled but not randomized = 28; Randomized = 608; Intent to treat = Randomized and received at least 1 dose. Events presented below from Randomized population, treatment-emergent (ITT).
Arm/Group | Placebo | Pramlintide 360 mcg | Metreleptin 5.0 mg | Pramlintide 180 mcg + Metreleptin 2.5 mg | Pramlintide 180 mcg + Metreleptin 5.0 mg | Pramlintide 360 mcg + Metreleptin 1.25 mg | Pramlintide 360 mcg + Metreleptin 2.5 mg | Pramlintide 360 mcg + Metreleptin 5.0 mg
Serious Adverse Events (participants affected / at risk) | 3/75 | 1/77 | 0/72 | 2/75 | 0/78 | 0/78 | 0/78 | 2/75
Other Adverse Events (participants affected / at risk) | 60/75 | 66/77 | 63/72 | 67/75 | 71/78 | 68/78 | 72/78 | 68/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=75) | Pramlintide 360 mcg (N=77) | Metreleptin 5.0 mg (N=72) | Pramlintide 180 mcg + Metreleptin 2.5 mg (N=75) | Pramlintide 180 mcg + Metreleptin 5.0 mg (N=78) | Pramlintide 360 mcg + Metreleptin 1.25 mg (N=78) | Pramlintide 360 mcg + Metreleptin 2.5 mg (N=78) | Pramlintide 360 mcg + Metreleptin 5.0 mg (N=75)
Food Allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope vasovagal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parathyroid Tumor benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Goiter (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=75) | Pramlintide 360 mcg (N=77) | Metreleptin 5.0 mg (N=72) | Pramlintide 180 mcg + Metreleptin 2.5 mg (N=75) | Pramlintide 180 mcg + Metreleptin 5.0 mg (N=78) | Pramlintide 360 mcg + Metreleptin 1.25 mg (N=78) | Pramlintide 360 mcg + Metreleptin 2.5 mg (N=78) | Pramlintide 360 mcg + Metreleptin 5.0 mg (N=75)
nausea (Gastrointestinal disorders) | 4 (4) | 31 (37) | 4 (4) | 27 (30) | 21 (22) | 26 (27) | 29 (32) | 19 (20)
injection site erythema (General disorders) | 1 (1) | 7 (8) | 15 (25) | 15 (17) | 17 (21) | 8 (9) | 24 (25) | 21 (24)
injection site pruritus (General disorders) | 1 (1) | 4 (4) | 13 (19) | 19 (20) | 21 (23) | 11 (11) | 18 (20) | 22 (23)
injection site bruising (General disorders) | 11 (14) | 11 (13) | 9 (13) | 9 (16) | 9 (9) | 11 (13) | 8 (9) | 16 (23)
injection site hemorrhage (General disorders) | 3 (3) | 10 (11) | 13 (17) | 14 (17) | 10 (10) | 7 (7) | 10 (11) | 11 (12)
injection site urticaria (General disorders) | 0 (0) | 2 (2) | 12 (12) | 13 (13) | 12 (12) | 5 (5) | 11 (14) | 11 (11)
Upper respiratory tract infection (Infections and infestations) | 8 (9) | 8 (9) | 2 (2) | 7 (7) | 10 (10) | 11 (11) | 9 (13) | 5 (5)
injection site rash (General disorders) | 0 (0) | 2 (2) | 13 (15) | 3 (5) | 8 (9) | 9 (12) | 12 (12) | 7 (10)
nasopharyngitis (Infections and infestations) | 4 (5) | 8 (9) | 8 (11) | 3 (5) | 4 (5) | 6 (9) | 6 (7) | 4 (7)
injection site nodule (General disorders) | 3 (3) | 2 (2) | 8 (11) | 3 (3) | 10 (10) | 2 (2) | 6 (6) | 8 (10)
headache (Nervous system disorders) | 4 (4) | 5 (5) | 4 (5) | 3 (3) | 7 (13) | 3 (3) | 3 (3) | 4 (4)
diarrhea (Gastrointestinal disorders) | 5 (5) | 5 (5) | 3 (3) | 5 (5) | 4 (4) | 4 (5) | 7 (7) | 3 (3)
urinary tract infection (Infections and infestations) | 5 (6) | 7 (13) | 3 (3) | 2 (2) | 2 (2) | 3 (5) | 3 (3) | 1 (1)
blood creatine phosphokinase increased (Investigations) | 6 (6) | 2 (2) | 1 (1) | 4 (4) | 3 (3) | 1 (2) | 5 (5) | 1 (1)
injection site induration (General disorders) | 3 (3) | 2 (2) | 2 (4) | 0 (0) | 6 (7) | 2 (2) | 1 (1) | 5 (5)
injection site inflammation (General disorders) | 0 (0) | 0 (0) | 1 (4) | 3 (3) | 4 (4) | 3 (3) | 3 (4) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 2 (2) | 3 (3) | 3 (4)
fatigue (General disorders) | 1 (1) | 3 (3) | 3 (3) | 5 (5) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
gastroenteritis viral (Infections and infestations) | 2 (2) | 4 (5) | 2 (2) | 3 (3) | 3 (3) | 1 (1) | 1 (1) | 2 (2)
constipation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2) | 5 (5) | 3 (3) | 2 (2) | 0 (0) | 2 (2)
vomiting (Gastrointestinal disorders) | 0 (0) | 6 (6) | 3 (3) | 0 (0) | 2 (2) | 5 (5) | 1 (1) | 1 (1)
dizziness (Nervous system disorders) | 4 (4) | 3 (3) | 1 (1) | 4 (4) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1) | 4 (4) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 2 (2) | 3 (3) | 0 (0)
sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
sinusitis (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 1 (1) | 2 (3) | 2 (2) | 4 (4) | 5 (5) | 5 (5) | 2 (2)

LIMITATIONS AND CAVEATS:
Drug Randomization stratified:sex,3 categories baseline BMI (12 arms); 3 treatment arms combined for summaries as single placebo treatment group; 3 combined for summaries as single pramlintide monotherapy treatment group (total:8 treatment groups).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.